CLINICAL TRIAL: NCT04280237
Title: Pharmacological Study of Cefazolin Antibioprophylaxis in Liver Transplantation
Acronym: ProCeTH
Status: Withdrawn | Type: Observational
Why Stopped: abandoned project
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI20/ProCeTH; 2020-A00405-34 (Other: IdRCB)
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Liver Transplant Infection; Surgical Site Infection; Antibiotic Prophylaxis; Cephazolin Adverse Reaction
Keywords: antibiotic prophylaxis; liver transplant; surgical site infection; Cefazolin
MeSH Terms: conditions — Surgical Wound Infection | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cefazolin in liver transplantation: Patient undergoing liver transplant surgery and receiving antibiotic prophylaxis with Cefazolin
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Blood samples

SUMMARY:
This study describes Cefazolin pharmacokinetics variation to target levels during liver transplantation.

DETAILED DESCRIPTION:
Cefazolin is one of the many drugs used in antibiotic prophylaxis during liver transplantation. However there are no study describing its pharmacokinetics during liver transplantation.

Due to the severe pharmacokinetics interactions caused by both prior hepatopathy and surgical techniques we suppose that Cefazolin blood levels are very different from those targeted for antibiotic prophylaxis.

This study aim to describe pharmacokinetics of Cefazolin during liver transplantation in order to adapt antibiotic prophylaxis strategy in case of unadapted measured levels.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* patient undergoing liver transplantation
* receiving Cefazolin as perioperative antibiotic prophylaxis to prevent surgical site infections

Exclusion Criteria:

* pregnant women
* legal protection or protected adults
* ongoing antibiotic treatment before liver transplantation
* patient inability to receive information or express opposition to the study.
* patient refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient receiving Cefazolin as perioperative antibiotic prophylaxis during liver transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Cefazolin blood concentration | Baseline up to 10 hours
  Cefazolin blood concentration will be measured at the moment of surgical incision and every hour until end of surgery

SECONDARY OUTCOMES:
Assess correlations between Cefazolin blood concentration and CHILD-PUGH score | baseline
  Patient's CHILD-PUGH score before transplantation
Assess correlations between Cefazolin blood concentration and MELD score | baseline
  Patient's MELD score before transplantation
Assess correlations between Cefazolin blood concentration and Cirrhosis etiology | baseline
  Cause of cirrhosis
Assess correlations between Cefazolin blood concentration and Transplantation indication | baseline
  Cause leading to transplantation
Assess correlations between Cefazolin blood concentration and Transjugular intrahepatic portosystemic shunt (TIPS) | baseline
  Medical history of TIPS
Assess correlations between Cefazolin blood concentration and Creatinine | baseline
  Creatinine levels will be measured before transplantation
Assess correlations between Cefazolin blood concentration and Hemodialysis | baseline
  Patient needing hemodialysis before liver transplantation
Assess correlations between Cefazolin blood concentration and Albumin | baseline
  Albumin levels will be measured before transplantation
Assess correlations between Cefazolin blood concentration and Surgery duration | End of surgery
  Time of surgical incision and end of the surgery will be noted
Assess correlations between Cefazolin blood concentration and Portal vein clamping time | End of surgery
  Time of portal vein clamping and declamping during realization of vascular anastomosis will be noted
Assess correlations between Cefazolin blood concentration and Ascitis | Baseline
  Volume of ascitis drained at the beginning of surgery
Assess correlations between Cefazolin blood concentration and Urine output | End of surgery
  Volume of urine output during surgery
Assess correlations between Cefazolin blood concentration and Blood loss | End of surgery
  Blood loss quantification will be done throughout surgery
Assess correlations between Cefazolin blood concentration and Red cell transfusion unit | End of surgery
  The number of red cell units transfused during transplantation will be counted at the end of surgery
Assess correlations between Cefazolin blood concentration and Platelet transfusion unit | End of surgery
  The number of platelet units transfused during transplantation will be counted at the end of surgery
Assess correlations between Cefazolin blood concentration and Plasma transfusion unit | End of surgery
  The number of plasma units transfused during transplantation will be counted at the end of surgery
Assess correlations between Cefazolin blood concentration and Intraoperative blood salvage | End of surgery
  Intraoperative blood salvage transfusion volume during surgery
Assess correlations between Cefazolin blood concentration and Crystalloid infusion | End of surgery
  Assess correlations between Cefazolin blood concentration and Volume of crystalloid infusion during surgery
Assess correlations between Cefazolin blood concentration and Colloid infusion | End of surgery
  Volume of colloid infusion during surgery
Assess correlations between Cefazolin blood concentration and Basal cardiac index | Baseline
  Cardiac index value at the beginning of surgery
Assess correlations between Cefazolin blood concentration and Minimal cardiac index | End of surgery
  Minimal index value during surgery
Assess correlations between Cefazolin blood concentration and Surgical site infection | Day 28
  Number of patient with surgical site infection in the 28 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Charlotte TELLIER, MD, Principal Investigator — University Hospital, Tours
Locations (1):
- Surgical intensive care unit, University Hospital, Tours, Tours, France